CLINICAL TRIAL: NCT05244603
Title: Application of Ideal Binary Masking to Disordered Speech
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Responsible Party: Principal Investigator, Sarah Leopold, Primary Investigator, Utah State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 10710
Record Dates: First submitted 2022-02-04; First posted 2022-02-17 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Hearing Loss, Sensorineural; Dysarthria
MeSH Terms: conditions — Hearing Loss, Sensorineural; Dysarthria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Hearing (Experimental): Listeners with normal hearing
  Interventions: Behavioral: Ideal binary mask
- Hearing Impaired (Experimental): Listeners with hearing loss
  Interventions: Behavioral: Ideal binary mask

INTERVENTIONS:
Behavioral: Ideal binary mask — Speech in noise processed by ideal binary mask to reduce background noise

SUMMARY:
Dysarthria and hearing loss are communication disorders that can substantially reduce intelligibility of speech and the addition of background noise adds a further challenge. This proposal utilizes an established signal processing technique, currently exploited for improved understanding of speech in noise for listeners with hearing loss, to investigate its potential application to overcome speech-in-noise difficulties for listeners understanding dysarthric speech. Successful completion of this project will demonstrate proof-of-concept for the application of this signal processing technique to dysarthric speech in noise, and inform the development of an R01 proposal to perform a large-scale evaluation of the technology, and clinically meaningful implications, in a broad range of disordered speech types and severities.

ELIGIBILITY:
Inclusion Criteria:INCLUSION CRITERIA for All Participants

* Native speakers of American English
* No history of speech or language impairment
* No significant prior contact with persons having neurogenic speech disorders

INCLUSION CRITERIA for Participants with Normal Hearing

* 18 to 70 years of age
* Auditory thresholds of 20 dB HL or better bilaterally at octave frequencies from 250-8000 Hz (if under 55 years of age)
* Auditory thresholds of 25 dB HL or better bilaterally at octave frequencies from 250-4000 Hz (if over 55 years of age)

INCLUSION CRITERIA for Participants with Sensorineural Hearing Loss

* 18 to 90 years of age

Exclusion Criteria:

* EXCLUSION CRITERIA for All Participants
* Mild or profound hearing loss
* Conductive or mixed hearing loss
* Asymmetric hearing loss
* Obvious concomitant cognitive or mental impairment
* Unable to achieve upward of 20% words correct

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Utah State University, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Borrie SA, Yoho SE, Healy EW, Barrett TS. The Application of Time-Frequency Masking To Improve Intelligibility of Dysarthric Speech in Background Noise. J Speech Lang Hear Res. 2023 May 9;66(5):1853-1866. doi: 10.1044/2023_JSLHR-22-00558. Epub 2023 Mar 21. PMID 36944186

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal Hearing | Hearing Impaired
Started | 422 | 13
Completed | 422 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Hearing | Hearing Impaired | Total
Number analyzed (Participants) | 422 | 13 | 435
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 410 | 4 | 414
  >=65 years | 12 | 9 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Overall represents both groups of listeners, row populations are subgroups
  years | 35 (12) | 69 (26) | 52 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204 | 7 | 211
  Male | 218 | 6 | 224
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 0 | 31
  Not Hispanic or Latino | 391 | 13 | 404
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 0 | 4
  Asian | 31 | 0 | 31
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 0 | 19
  White | 363 | 13 | 376
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 422 | 13 | 435
Speech intelligibility +5 dB SNR [Mean (Standard Deviation); unit: percentage of words correct] — Population: Overall represents both groups of listeners, row population represents subgroups
  percentage of words correct | 40 (5) | 24 (16) | 32.5 (10.5)

OUTCOME MEASURES:

1. Primary Outcome: Percent Correct Speech Intelligibility
Description: Percent of keywords correctly identified by the participant for the processed speech stimuli, listeners were presented with phrases containing several words and they reported back what they heard. The number of words corrected reported by each listener was counted and converted to a 'percent correct' score.
Time Frame: One hour
Population: Listeners with normal hearing and listeners with hearing loss
Measure: Mean (Standard Error); unit: percentage of words correctly reported
Arm/Group | Normal Hearing | Hearing Impaired
Number analyzed (Participants) | 422 | 13
percentage of words correctly reported | 69 (1.06) | 63 (2.2)

ADVERSE EVENTS:
Time Frame: 2 years 29 days
Arm/Group | Normal Hearing | Hearing Impaired
All-Cause Mortality (participants affected / at risk) | 0/422 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/422 | 0/13
Other Adverse Events (participants affected / at risk) | 0/422 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT05244603/Prot_SAP_ICF_000.pdf